CLINICAL TRIAL: NCT03903289
Title: Assessment of Implementation of the Automated Erythrocytapheresis in the Outcome of Egyptian Sickle Cell Disease Patients: Single Center Experience
Brief Title: The Implementation of the Automated Erythrocytapheresis in Egyptian Sickle Cell Disease Center
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Fatma Soliman Elsayed Ebeid, MD, Assistant Professor of Pediatric, Ain Shams University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU M D 94/ 2018
Record Dates: First submitted 2019-03-14; First posted 2019-04-04 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Automated red cell exchange (Experimental): Automated red cell exchange
  Interventions: Procedure: Automated red cell exchange
- Manual red cell exchange (Active Comparator): Manual red cell exchange
  Interventions: Procedure: Manual red cell exchange
- Simple red cell transfusion (Sham Comparator): Simple red cell transfusion
  Interventions: Procedure: Simple red cell transfusion

INTERVENTIONS:
Procedure: Automated red cell exchange — Erythrocytapheresis is an automated red cell exchange procedure that removes blood that contains HbS from the patient while simultaneously replacing that same volume with packed red cells free of HbS.
  Other Names: Erythrocytapheresis
  Arms: Automated red cell exchange
Procedure: Manual red cell exchange — Active Comparator: Manual red cell exchange
  Arms: Manual red cell exchange
Procedure: Simple red cell transfusion — Active Comparator: Simple red cell transfusion
  Arms: Simple red cell transfusion

SUMMARY:
Improvements of health infrastructure, preventive care and clinical treatment have reduced the morbidity and mortality of sickle cell disease (SCD). However, SCD is still an increasing national health problem, with increase longevity the chronic effect of sustained hemolysis and episodic vaso-occlusive events and the recurrent episodes of ischemic reperfusion injury drive the development of progressive end organ complications and cardiovascular, pulmonary, neurological and renal systems are most commonly affected. Today there is hope for a cure using hematopoietic stem cell transplantation (HSCT). However, at present; the procedure is infrequently performed and very expensive. In this research we will assess the effect of implementation of the automated erythrocytapheresis in the outcome of sickle cell disease in single Egyptian center.

DETAILED DESCRIPTION:
There is a wide scoop for treatment of SCD ranging from medical treatment with hydroxyurea, simple transfusion with chelation therapy, exchange transfusion either manual or automated and stem cell transplantation which need highly equipped institutes.

The goals of treatment of SCD are symptom control with early detection and management of disease complications. Although several pharmacological agents have been studied for the treatment of SCD, the only drug currently approved by the US Food and Drug Administration (FDA) for the treatment of SCD is hydroxyurea. Allogeneic bone marrow transplantation (BMT) can cure SCD, but it is difficult to decide which patients should be offered BMT. Many risks are associated with BMT, and the risk-to-benefit ratio must be assessed carefully. The lack of availability of a matched donor may limit the utility of BMT. Transfusions are not needed for the usual anemia or episodes of pain associated with SCD. Urgent replacement of blood is often required for sudden severe anemia and regular blood transfusions are used for primary and secondary stroke prevention in children with SCD. With continued transfusion, iron overload inevitably develops and can result in heart and liver failure, and multiple other complications necessitate the use of chelation therapy.

Erythrocytapheresis is an automated red cell exchange procedure that removes blood that contains HbS from the patient while simultaneously replacing that same volume with packed red cells free of HbS. Transfusion usually consists of sickle-negative, leuco-reduced, and phenotypically matched blood for red cell antigens. Erythrocytapheresis thus has the advantage of controlling iron accumulation in patients with SCD who undergo long-term transfusion, as well as the ability to allow rapid reduction of HbS concentrations to less than 30% without significantly increasing total hemoglobin concentration post transfusion. This precision is achieved because, before the start of the transfusion, the computer in the pheresis machine calculates the expected amount of packed RBCs required to obtain a specific post-transfusion hemoglobin level, using various physiologic parameters (eg, height, weight, Hb level). Further, erythrocytapheresis requires less time than simple transfusion of similar blood volumes. Although erythrocytapheresis is more expensive than simple transfusion, the additional costs associated with simple transfusions (ie, those of chelation and organ damage due to iron overload) make erythrocytapheresis more cost-effective than simple transfusion programs. Central venous access devices can safely be used for long-term erythrocytapheresis in patients with SCD with a low rate of complications.

ELIGIBILITY:
Inclusion Criteria:

* Patient with sickle cell disease (HbS with other variant hemoglobin)
* Age from 2-30y old

Exclusion Criteria:

Patients with other hemoglobinopathy Patients younger than two years

Ages: 2 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-08-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
The change of health related quality of life (HRQoL) is being assessed | assessed at enrollment and after one year of intervention
  The medical Outcome Study (MOS) short form (SF-36) is a 36- item tool for measuring health status and outcome from the patients' perceptions

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Solima SE Ebeid, MD, Principal Investigator — Faculty of Medicine, Ain Shams university
Locations (1):
- Faculty of Medicine, Ain Shams University, Cairo, Non-US, Egypt